CLINICAL TRIAL: NCT05596305
Title: Outcomes of Anti Stigma Educational Intervention of Undergraduate Medical Students Towards Mentally Ill Patients-Suez Canal University Hospital
Brief Title: Outcomes of Anti Stigma Educational Intervention of Ungraduated Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Ismail Dahshan, senior lecturer family medicine, Suez Canal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1772018AntiStigMed
Record Dates: First submitted 2022-09-18; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Stigmatization; Medical Education
MeSH Terms: conditions — Stereotyping

STUDY DESIGN:
Intervention Model Description: quasi experimental ( pre-post ) study evaluating the outcomes of anti-stigma educational intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- undergraduate medical students (Experimental): an educational anti-stigma intervention delivered to undergraduate medical students comparing the outcomes of the study before and after the intervention at two time intervals
  Interventions: Behavioral: educational psychiatry intervention

INTERVENTIONS:
Behavioral: educational psychiatry intervention — educational anti-stigma intervention related to psychiatric illness composed of a lecture, video, role models play, and open discussion

SUMMARY:
Background: Stigma causes a significant burden for mental ill patients. Unfortunately, negative attitudes towards mentally ill are not confined to the lay public but are also common among health professionals.

Aim: To study outcomes of psychiatric anti stigma educational intervention on undergraduate medical students' knowledge, attitude, and behavior as primary outcome measures.

Subjects and methods: a quasi-experimental study was conducted on fourth year (120) undergraduate medical students affiliated to faculty of Medicine-Suez Canal University. The participants conducted a semi-structured questionnaire to assess effect of anti-stigma program on their knowledge, attitude and intended behavior toward mentally ill. The participants completed baseline questionnaire, then immediately and after 6 months reassessment. Data was collected from November 2019 to May 2020.

DETAILED DESCRIPTION:
Subjects and Methods:

The current study was a quasi-experimental (pre-post) intervention study was conducted on 120 all fourth-year undergraduate medical students affiliated to faculty of medicine, Suez Canal University in Ismailia city, Egypt to assess the outcomes of psychiatric anti-stigma educational intervention on their knowledge, attitude and intended behavior toward mentally ill. Permissions for the study were obtained from the authorities concerned, and the participants medical students were informed about the purpose of the study and signed an informed consent before the beginning of this study.

Methods:

The First part: Consists of socio-demographic data of each medical student, which includes age, gender, family history of mental illness and contact with mentally ill patients in the past 3 months and if he/she received the previous year's seminars or workshops related to the stigma of mental illness.

The second part: Consists of Specific items that measure mental health-related knowledge among the general public using the Mental Health Knowledge Schedule (MAKS), its validity is supported by extensive review by experts including service users and international experts in stigma research and has been found to be brief and feasible with internal reliability and test-retest reliability moderate to substantial [11].. Part A of the scale comprises six items covering stigma-related mental health knowledge areas (need for paid employment, advice for professional help, medication is effective, psychotherapy is effective, full recovery from mental illness, seeking professional help by mentally ill) and Part B consists of six items that inquire about the classification of various conditions as mental illnesses to help contextualize the responses to other items. A 5-point Likert scale was used, and response options range from 1 = totally disagree to 5 = totally agree. "Don't know" was valued at 3 for the purposes of determining a total score. Items 6, 8 and 12 are reverse coded to reflect the direction of the correct response. The total score was calculated by adding the response values for only items 1-6 (Part A) and ranged from 6 to 30. A higher score indicates more knowledge. The Cronbach's alpha for the MAKS scale was 0.749.

The third part: Used, the Beliefs towards Mental Illness scale (BMI) to assess the attitudes toward mental illness, the scale was designed to measure cross-cultural differences in such beliefs as well as to predict treatment-seeking behavior among different cultural groups, with reliability estimates for each factor revealed to be moderate to high internal consistency [12]. It is composed of 21 items that measure negative stereotypical views of mental illness. The BMI scale consists of three subscales; Dangerousness subscale: Consists of five items (1, 2, 3, 6, 13) relating to the perceived dangerousness of mental illness and patients; Social and interpersonal skills subscale: Consists of 10 items (4, 5, 8, 11, 12, 14, 15, 17, 18, 21) covering the effect of mental illness on interpersonal relationships and related feelings of despair. It assesses the level of frustration and despair in interpersonal relationships with individuals with a mental illness. Also, taps feelings of shame about mental illness and the perception that the mentally ill are untrustworthy; and Incurability subscale: Consists of six items (7, 9, 10, 16, 19, 20) covering perceptiveness of incurability of mental illness. Items are rated on a five-point Likert scale, reverse coded from 1 (strongly agreement) to 5(strongly disagree). The total score was calculated by adding the response values for 21 items and ranged from 21 to 105. The lower score reflects a more negative belief toward the mentally ill. The Cronbach's alpha for the BMI scale was 0.82 and the subscales were between 0.69 - 0.80.

The fourth part: Assesses the mental health-related reported and intended Behavior measured by the Reported and Intended Behavior Scale (RIBS), Which was found to be a brief, feasible and psychometrically robust measure for assessing health-related reported and intended behavioral discrimination, with moderate to substantial internal consistency and test-retest reliability [13]. The four reported behavior outcomes included, living with, working with, living nearby, and continuing a relationship with someone with a mental health problem, while the four-intended behavior outcomes assessed the future intended behavior of the same items. A 5-point Likert scale was used, and response options range from 1 = totally disagree to 5 = totally agree. "Don't know" was valued at 3 for the purposes of determining a total score. The total score for each student is calculated by adding together the response values for intended behavior items and ranges from 4 to 20. A higher score indicates more favorable intended behavior. The Cronbach's alpha for the RIBS scale was 0.75. Ethical approval for carrying out the study was obtained from The Ethical Committee of the Faculty of Medicine, Suez Canal University, and the participant students were informed about the purpose of the study and signed informed consent before the start of the study.

Intervention program:

This study was carried from September 2019 to February 2020. Educational non discriminative anti-stigma educational intervention was delivered before the formal psychiatry rotation in the fourth year of the undergraduate study, and participation was voluntary. the intervention consisted of a 2-hour interactive lecture which explained the key facts and figures about stigma and discrimination related to mental illness, causes and consequence of stigma, video showed examples of social stigma related to mental illness and its impact on mental ill patients and their family, and how to combat stigma related to mental illness and ended by open discussion with students for any questions. Subsequently, half an hour personal testimony about the experience of mental health problems and stigma from person with direct experience of schizophrenia after his recovery, using trained role-player who had some theatre experiences. Then followed by, half an hour role-plays in small groups, using trained role-players to act the part of service users who suffer from depression and caregiver of schizophrenic patient.

Statistical analysis:

The data of the current study were analyzed using the SPSS version 20 (i.e., statistical package for social sciences) program. According to the results of the Shapiro-Wilk test for normality, continuous data were expressed as the median and interquartile range (IQR). Spearman correlation coefficient test was conducted to find the correlation between medical students' knowledge, attitude and behavior, toward mentally ill patients and different demographic variables. The scores of mental health-related knowledge, belief towards mental illness (with its 3 subscales), and intended behavior were categorized as poor or good based on the threshold score (cut-off point) obtained from the Likert scale which is ordinal but is often analyzed as numerical neglecting the differences between ordinal scores according to the following formula: The threshold score = ([total highest score-total lowest score]/2) + total lowest score. Predictors of baseline knowledge, belief, and behavior scores were determined using univariate linear regression analysis. If more than one significant predictor existed, the significant variables were implemented in a multivariate regression analysis. After accomplishment of the educational program, comparison of the knowledge, belief, and behavior scores across time was done using Related-Samples Friedman's Two-Way Analysis of Variance by Ranks. Pairwise analysis was performed to assess the difference between each two time periods. Males and females were compared concerning the studied scores using Mann-Whitney test. P values less than 0.05 were considered significant. The results were presented as tables, and graphs.

ELIGIBILITY:
Inclusion Criteria:

* All fourth-year medical students in the faculty of medicine, Suez Canal University.

Exclusion Criteria:

* Refusal to participate and/or decline to complete the study for any cause.
* Any Identified history or treatment for psychiatric conditions.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-11-03 (Actual); Primary Completion 2020-05-17 (Actual); Study Completion 2020-05-17 (Actual)

PRIMARY OUTCOMES:
The cut-off point score of MAKS assessed at the baseline, immediately after the intervention, and at 6-months follow up. | 0-6 months
  The Mental Health Knowledge Schedule (MAKS). It is a 5-point Likert scale ranging from 6 to 30, and the higher score indicates more mental health knowledge.
The cut-off point score of BMI assessed at the baseline, immediately after the intervention, and at 6-months follow up. | 0-6 months
  The Beliefs toward Mental Illness scale (BMI) consists of 3 subscales measuring dangerousness, Social and Interpersonal skills, and incurability. BMI is a 5-point Likert scale, consists of total 21 items, and ranging from 21 to 105. The higher score indicates more favorable beliefs towards mental illnesses
The cut-off point score of RIBS assessed at the bassline, immediately after the intervention, and at 6- months follow up. | 0-6 months
  RIBS is a 5-points Likert scale, ranging from 4 to 20 with higher score indicates more favorable intended behavior with mentally ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Dahshan, PhD, Principal Investigator — Suez Canal University
Locations (1):
- Faculty of medicine , Suez Canal University, Ismailia, Egypt